CLINICAL TRIAL: NCT00206713
Title: Phase 3 Randomized, Double-Blind, Placebo-Controlled Multicenter Retreatment Study of Sargramostim (Leukine®) in Patients With Active Crohn's Disease and Prior Treatment Response to Sargramostim
Brief Title: Efficacy Study of Sargramostim in the Retreatment of Patients Who Have Crohn's Disease Who Have Previously Responded to Treatment With Sargramostim
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 308180; 91404; Novel 3
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Crohn Disease
Keywords: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — sargramostim

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Sargramostim (Leukine)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sargramostim (Leukine) — 6 μg/kg sargramostim administered SC once daily for 8 weeks
  Other Names: BAY86-5326
  Arms: Arm 1
Drug: Placebo — Placebo administered SC once daily during the randomized retreatment phase.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate whether treatment with Leukine in patients with Crohn's disease who have previously responded to Leukine can be helped again, once they have relapsed.

DETAILED DESCRIPTION:
On 29 May 2009, Bayer began transitioning the sponsorship of this trial to Genzyme. NOTE: This study was originally posted by sponsor Berlex, Inc. Berlex, Inc. was renamed to Bayer HealthCare, Inc.

ELIGIBILITY:
Inclusion Criteria:

* You must be 18 years or older.
* You must have active Crohn's disease at the time of screening.
* You must be 18 years or older.
* You must have active Crohn's disease at the time of screening.
* You must be able to give yourself an injection of study drug or have another person who can help you give the injection.
* You must not be pregnant and agree to use birth control if you are a sexually active male or female of childbearing potential.

Exclusion Criteria:

* You may not be pregnant or breastfeeding.
* You may not have a colostomy or ileostomy.
* You may not be taking prohibited medications.
* You may not have had GI surgery or a bowel obstruction in the last 6 months.
* You may not have ever taken this drug or drugs of similar type in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2004-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving clinical response or remission | At Day 57 of the randomized retreatment phase

SECONDARY OUTCOMES:
Proportion of patients achieving clinical response or remission | At the end of Week 8 of the open-label phase.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (7):
- United States (7):
  - San Francisco, California
  - Atlanta, Georgia
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Morristown, New Jersey
  - Philadelphia, Pennsylvania
  - Houston, Texas